CLINICAL TRIAL: NCT06128200
Title: Randomized Controlled Trial Comparing NEUROMARK System to Sham Control in Patients With Chronic Rhinitis
Brief Title: NEUROMARK Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurent Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CIP-0010
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Chronic Rhinitis

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized, sham-controlled, single-blinded, superiority trial
Who Masked: Participant
Masking Description: This is a single-blind study; participants will be blinded to the randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active (Active Comparator): Subjects in this arm will undergo treatment with the NEUROMARK device.
  Interventions: Device: NEUROMARK System
- Sham (Sham Comparator): Subjects in this arm will undergo the procedure with a Sham device. Sham control participants will be offered the option to receive active treatment after the 90-day follow-up provided they still meet all eligibility criteria.
  Interventions: Device: Sham NEUROMARK System

INTERVENTIONS:
Device: NEUROMARK System — The NEUROMARK System is indicated for use in otorhinolaryngology (ENT) surgery for creation of radiofrequency (RF) lesions to disrupt posterior nasal nerves in patients with chronic rhinitis.
  Arms: Active
Device: Sham NEUROMARK System — Sham ablation procedure using the NEUROMARK System
  Arms: Sham

SUMMARY:
The NEUROMARK RCT Study is a prospective, multicenter, randomized, sham-controlled, single-blinded, superiority trial.

ELIGIBILITY:
Inclusion Criteria:

Participant Must:

1. Be ≥18 years of age.
2. Have been experiencing rhinitis symptoms for a minimum of 6 months.
3. Have moderate to severe symptoms of runny nose (individual rTNSS symptom rating of 2 or 3), mild to severe symptoms of nasal congestion (individual rTNSS symptom rating of 1,2, or 3), and a minimum total score of 5 (out of 12) at baseline.
4. Be an appropriate candidate for bilateral NEUROMARK device treatment performed under local anesthesia.
5. Be willing and able to comply with all study elements, as indicated by written informed consent.

Primary Exclusion Criteria:

Participant Must Not:

1. Have clinically significant anatomic obstruction that in the investigator's opinion limit access to the posterior nose, including but not limited to severe septal deviation or perforation, nasal polyps, and/or sinonasal tumor.
2. Have had previous sinus or nasal surgery within 6 months of study enrollment.
3. Have previously undergone RF, cryotherapy, or other surgical interventions for rhinitis.
4. Have rhinitis symptoms that are due to seasonal allergies only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
rTNSS | 90-days post procedure follow-up
  Comparison of the percentage of responders (participants with a 30% or greater reduction in rTNSS relative to baseline) between study arms at 90-days

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - ExcelENT, Homewood, Alabama
  - East Alabama ENT, Opelika, Alabama
  - Sensa Health, Los Angeles, California
  - Sacramento ENT, Sacramento, California
  - Breathe Clear Institute, Torrance, California
  - ENT & Allergy Associates of Florida, Boynton Beach, Florida
  - ENT & Allergy Associates of Florida, Port Saint Lucie, Florida
  - Ascension St. Vincent, Anderson, Indiana
  - Kentuckiana, Louisville, Kentucky
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Centers for Advanced ENT Care, Baltimore, Maryland
  - Bethlehem ENT, Bethlehem, Pennsylvania
  - Houston Methodist ENT Specialists, Houston, Texas
  - The ENT & Allergy Centers of Texas, McKinney, Texas
  - Richmond ENT, Richmond, Virginia
  - ENT & Allergy Associates, Puyallup, Washington

IPD SHARING:
Plan to Share IPD: No